CLINICAL TRIAL: NCT01162083
Title: Identifying the Ideal Parameter of the Cardiopulmonary Exercise Test to Distinguish Between the Cardiovascular and Respiratory Components of Functional Limitation and to Detect Relevant Physiological Changes in Function
Brief Title: Identifying an Ideal Cardiopulmonary Exercise Test Parameter
Acronym: PVA
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Humboldt-Universität zu Berlin (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CRO1570
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2011-08

CONDITIONS: Left Ventricular Systolic Dysfunction; Mitral Regurgitation
Keywords: Exercise Physiology; Cardiopulmonary Interaction; Heart Failure
MeSH Terms: conditions — Ventricular Dysfunction, Left; Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Mitral Valve disease: Patients with mitral valve disease, deemed suitable and ready for elective valve repair or replacement. No significant arrhythmias, other valvular disease or LV dysfunction present. We shall also be recruiting patients undergoing a Mitraclip procedure.
- COPD: Patients with isolated chronic obstructive pulmonary disease and no cardiac disease.
- Mixed Lesions: Patients with proven limitation from both cardiac and respiratory disease.
- CRT: Patients with symptomatic heart failure who have responded to cardiac resynchronisation therapy (biventricular pacemaker).
- Cardiomyopathy: Heart Failure of primarily myopathic origin, without rhythm disturbance, ongoing ischaemia or significant valvular disease.

SUMMARY:
Cardiopulmonary exercise testing (CPET) is a safe, noninvasive investigation where a patient walks on a treadmill or cycles whilst attached to an ECG and with a mask that measures the air breathed in and out. It has numerous clinical uses, such as diagnosing the main cause in patients with breathlessness, deciding on timing for heart transplantation and assessing whether patients are safe for a general anaesthetic.

A patient's peak oxygen consumption, the maximum amount of oxygen taken up by the blood from the lungs when breathing increases during exercise, is the main measurement taken from CPET. It is low in heart disease and has been used to predict the risk of death and therefore plan treatments for patients. However this is also low in numerous other diseases including lung disease; reduced oxygen consumption in patients with two conditions may be wrongly thought to be because of the heart leading to inappropriate action and distress to the patient.

Newer measurements of exercise capacity from the same exercise test are better at predicting death in heart failure.

We propose that they are more specific for heart failure over other diseases, for example lung disease, when compared with peak oxygen consumption, and are superior when a single best test for heart failure is required.

This research aims to identify which measurement of exercise capacity is most specific for heart failure. We will perform the test on many patients with different diseases, and before and after procedures such as the implantation of special pacemakers, and heart valve operations. This should lead to a more accepted use of this investigation and the more appropriate identification of which patient should have which procedure.

DETAILED DESCRIPTION:
Heart failure, where the heart muscle is damaged and is unable to pump blood efficiently, affects 9% of those aged 55 or more and is responsible for about 2% of the hospital admissions in the UK. The first symptom many patients complain of is breathlessness on exercise and an inability to perform their normal daily activities. Unfortunately these symptoms are similar to those experienced in numerous diseases of the heart and lungs. Cardiopulmonary exercise testing, through measuring numerous values taken from breathing during exercise can tell us which disease is causing the symptoms.

The leading parameter from a CPET, peak VO2, has for many years been the single value used to guide management of patients following a diagnosis of many diseases from the heart and lungs. Newer measures predict outcome from heart failure (our principal area of interest) better. We believe this may be because they are less affected by lung disease than peak VO2 and we know that many patients have both heart and lung diseases.

By showing the best CPET variable for each individual disease state, we will be able to ensure patients are correctly put into a level of risk for their condition and that they will be followed-up with the most accurate marker from exercise testing, rather than a "one size fits all" approach of peak VO2.

With regards to heart valve disease, standard exercise testing just using ECG leads, rather than cardiopulmonary exercise testing, is starting to be used more in identifying patients without symptoms for possible surgery. The inaccuracy of this test will inevitably lead to patients being wrongly categorised. Cardiopulmonary exercise testing is a much more accurate way of establishing the impact of any disease on the heart or lung over traditional exercise testing and therefore we believe that evidence of its role around the time of surgery could be used as further support for its role in improving decision making for patient.

Ultimately the greater knowledge of this test and when we should use it will help patients with very common heart conditions to be treated appropriately, potentially helping many patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years of age.
2. Able to perform cycle ergometry and agree to perform between 2 and 3 tests.
3. If previously undergone echocardiography there is evidence of reasonable echo windows (good views).
4. Agree to the full study protocol.

Exclusion Criteria:

1. Significant coexistent pathologies of the groups tested unless specifically in that group of mixed pathologies in the "Observational Study". This includes any combination of COPD or restrictive lung disease alongside heart failure and valvular disease. Therefore all cardiac conditions should have no significant limitation on spirometry, and all patients with lung disease should have good left ventricular function with no significant increases in pulmonary vascular pressures as seen on echocardiography. Patients with atrial fibrillation/ flutter will be excluded. Patients with more than mild valvular lesions will be excluded from all groups except the joint group and the group with mitral valvular disease
2. Symptomatic coronary disease, or significant ischaemia noted on cardiopulmonary exercise test (unless accounted for by aortic valve disease, in which case a prior coronary angiogram would have been undertaken if significant coronary disease then they will not be invited to participate).
3. Anaemia (Hb <12 in men, <11 in women).
4. Obesity (BMI >30) which could lead to limitation independent of the cardiovascular or respiratory condition.
5. Chronic Kidney Disease Stage 3 or above (estimated GFR <60ml/hr as calculated by Cockcroft Gault equation). The metabolic acidosis associated with this condition will affect ventilatory equivalents.
6. Poor echocardiographic windows so that a full data set is not achievable.
7. Inability to perform a symptom limited cardiopulmonary exercise test.
8. Inability to perform spirometry.
9. Inability to consent/make decisions (lack of competence)
10. Vulnerable adult/current detainee in prison/elsewhere.
11. Significant neurological or musculoskeletal abnormalities.
12. Inability to complete all the investigations at the time intervals agreed in the protocol.
13. Permanent Pacemaker unless in the biventricular pacemaker group in the Interventional Study. These patients in this group will be excluded if they are pacing dependent (when the biventricular function is disabled they do not have a normal intrinsic rhythm) and if they have significant first degree AV block at rest or on exercise (will activate right ventricular pacing after a sinus beat).
14. Patients in the atrial fibrillation interventional group will be excluded if they revert back to atrial fibrillation after the procedure, or the procedure never restores sinus rhythm. These patients will still be eligible for inclusion in the observational study.
15. Recent (recovery within <1month) decompensation of their underlying cardiac or respiratory disorder.
16. Uncontrolled hypertension.
17. Untreated life threatening arrhythmia.
18. Recent surgery (within 10 weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current patients under tertiary care for cardiac or respiratory disease. Valvular patients will be stable patients under follow-up to judge optimal timing for intervention on clinical grounds at which point they will become applicable to the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The relation or change between Cardiopulmonary exercise test variables | Up to 6 months
  In the Observational Cohort Study the primary outcome measure is the relation between variables (peak VO2, VE/VCO2, OUES, Tau, AT) when compared between the groups with different disease states.
  In the Interventional Cohort Study the primary outcome is the change in a variable (peak VO2, VE/VCO2, OUES, Tau, AT) from before to after an intervention which is required on clinical grounds.

SECONDARY OUTCOMES:
Using Cardiopulmonary Exercise Test Variables to help Assess for Functional Improvement | 6 months
  In patients undergoing heart valve replacements or an ablation for atrial fibrillation the improvement in symptomatic benefit will be compared to the change in cardiopulmonary exercise test variables.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Wensel, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Barron A, Francis DP, Mayet J, Ewert R, Obst A, Mason M, Elkin S, Hughes AD, Wensel R. Oxygen Uptake Efficiency Slope and Breathing Reserve, Not Anaerobic Threshold, Discriminate Between Patients With Cardiovascular Disease Over Chronic Obstructive Pulmonary Disease. JACC Heart Fail. 2016 Apr;4(4):252-61. doi: 10.1016/j.jchf.2015.11.003. Epub 2016 Feb 10. PMID 26874378